CLINICAL TRIAL: NCT01303328
Title: A Randomized, Double-blind, Multi-centre, Placebo Controlled Phase II Clinical Study to Evaluate the Efficacy, Tolerance and Safety of an Aqueous Gel Containing an Antiviral, Directly Applied on the Cervix Exhibiting High Grade Intraepithelial Lesion.
Brief Title: Safety and Efficacy Study of Antiviral Local Application to Treat High Grade Cervical Intraepithelial Lesions (CIN2/3)
Acronym: Colvir-PhaseII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mithra Pharmaceuticals (Industry)
Responsible Party: Maud Jost, Mithra Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CI-C02; 2010-023271-26 (EudraCT Number)
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2012-08

CONDITIONS: Uterine Cervical Neoplasia; Cervix Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: C1
- Placebo group (Placebo Comparator)
  Interventions: Drug: C1

INTERVENTIONS:
Drug: C1 — Local application of the experimental gel or placebo gel.

SUMMARY:
The purpose of this phase-II study is to evaluate the efficacy and safety of an aqueous gel containing an antiviral, administered directly on cervix exhibiting high grade squamous or glandular intraepithelial lesion (CIN 2 and 3) in comparison with a placebo treatment.

DETAILED DESCRIPTION:
Human Papilloma Virus (HPV) infections induce cervical intraepithelial neoplasia (CIN) of cervix. To reduce incidence of invasive tumor associated with high grade CIN lesions, the standard treatment is the conisation of cervix (surgical act). A local treatment with antiviral would preserve the cervix of young subjects and reduce obstetrical morbidity induced by the conisation.

This clinical study is aimed at:

* to evaluate the efficacy of a gel with antiviral directly applied on the cervix exhibiting high grade CIN lesions (CIN2/3): conisation is still indicated?
* to evaluate the safety and tolerance after local application.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 50 years old
* Informed consent signed
* Cervical lesion classified CIN 2 or 3, on a biopsy made during the 60 days before inclusion
* No sexual activity, or proved sterility, or use of effective mechanical, hormonal or intrauterine contraception during 30 days following inclusion (except vaginal ring Nuvaring, diaphragm and spermicide)

Exclusion Criteria:

* Invasive or microinvasive cervical neoplasia
* Pregnancy or breast feeding
* Subtotal hysterectomy
* Current renal impairment
* Current immune disorder including serology HIV +
* Current use of drugs interfering with renal function
* Current use of oncologic treatment
* Current use of immune treatment
* Current use of anti-viral treatment
* Current vaginal application of drugs or cosmetics
* Prior treatment with the antiviral on the cervix
* Local or general condition incompatible with the experimental treatment in the opinion of the principal investigator
* Current or recent participation to another experimental study during the last 3 months before the screening visit

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Efficacy at week 12: change of histological and cytological parameters (success or not) | 12 weeks
  Efficacy will be measured by histological and cytological criteria at week 12 (disappearance of CIN 2+) in correlation with viral status (positive or negative) before and after treatment.
Efficacy at week 28: recurrence rate | 28 weeks
  The recurrence rate will be assessed at week 28, by the same histological and cytological criteria in correlation with the viral status (positive or negative) before and after treatment.
Tolerance and Safety (AE reporting, changes of gynecological and biological parameters) | during 30 weeks
  Safety will be measured by record of adverse events, changes in clinical biology test results; local tolerance will be measured by patient questioning and gynecological examination of vagina and cervix.

SECONDARY OUTCOMES:
Virological status (infection) | during 30 weeks
  The viral load and genotypes of HPVhr will be determined before treatment, during follow-up and at the end of the study, by using a quantitative analysis.
Changes in lesion (colposcopic changes) | during 30 weeks
  Colposcopic description of lesion will be done before, during and after treatment of the lesion, during follow up and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe SIMON, MD, PhD, Professor, Principal Investigator — Hôpital Erasme, service de gynécologie obstétrique
Locations (9):
- Belgium (9):
  - Hôpital Saint Pierre, Brussels, Brussels Capital
  - CHU Brugmann, Brussels, Brussels Capital
  - Hôpital Erasme, Brussels, Brussels Capital
  - HIS Ixelles, Ixelles-Elsene, Brussels Capital
  - CHU Charleroi Hôpital Civil, Charleroi, Charleroi
  - CHU Charleroi Site André Vésale, Montigny-le-Tilleul, Charleroi
  - CHU Tivoli, La Louvière, La Louvière
  - CHU ND des Bruyères, Chênée, Liege
  - CHR Citadelle, Liège, Liege